CLINICAL TRIAL: NCT00664092
Title: Evaluating Alternative Aftercare Models for Ex-Offenders
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: DePaul University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Leonard Jason, Director Center for Community Research, DePaul University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: LJ070306PSY-C1; 5R01DA019935-03 (NIH)
Record Dates: First submitted 2008-04-18; First posted 2008-04-22 (Estimated); Last update posted 2015-02-11 (Estimated); Status verified 2015-02

CONDITIONS: Usual Aftercare; Oxford House; Therapeutic Community
Keywords: Substance Abuse; Ex-Offenders; Substance Abuse Recovery
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (No Intervention): Usual Aftercare Condition
- 2 (Experimental): Oxford House Condition
  Interventions: Other: Residential
- 3 (Experimental): Therapeutic Community Condition
  Interventions: Other: Residential

INTERVENTIONS:
Other: Residential — living in a democratic, resident-run setting
  Other Names: Oxford House
  Arms: 2
Other: Residential — Professionally-run substance abuse recovery setting
  Other Names: Safe Haven Therapeutic Community
  Arms: 3

SUMMARY:
The primary aim of this project is to study more closely the role played by post-release aftercare in the outcomes of criminal offenders who received in-prison substance abuse treatment. Prison-based therapeutic communities (TC) (Pelissier et al., 2001; Wexler, 1995) have demonstrated efficacy, especially when combined with post-release TC aftercare (Melnick et al., 2001). The aims of this project are important from a public health perspective as there may be treatment matching, case management, and financing factors that could be manipulated to enhance the cost-effectiveness of community-based substance abuse treatment for offenders leaving prison. It is possible that both TC and Oxford House(OH) aftercare modalities increase abstinence social support, self-efficacy, and employment, which mediate reductions in drug use, reincarceration, and health problems, but overall benefits are likely to be greater for TCs because they employ professional services and empirically based behavioral strategies. However, OHs might have advantages compared to more traditional post-incarceration modalities (e.g., low costs). Bringing scientific methods to the examination of TCs and the OH community-based recovery models for addiction might help to identify the "active ingredients" of these recovery settings.

DETAILED DESCRIPTION:
The primary aim of this project is to study more closely the role played by post-release aftercare in the outcomes of criminal offenders who received in-prison substance abuse treatment. Prison-based therapeutic communities (TC) (Pelissier et al., 2001; Wexler, 1995) have demonstrated efficacy, especially when combined with post-release TC aftercare (Melnick et al., 2001). For example, Inciardi et al. (2003) showed that TC aftercare substantially reduced criminal behavior and significantly decreased illicit drug use when compared to outcomes for inmates who dropped out of prison TC care or graduated prison TC, but who did not enter or remain long in TC aftercare. Moreover, some released TC participants may prefer and feel that they are ready for a less-structured environment than TC aftercare.

Several important questions relevant to public health issues remain unclear in the scientific literature regarding prison TC aftercare. The answers might help establish more enlightened post-release aftercare policy affecting prison inmates. For example, it is unclear whether the main therapeutic effect of TC aftercare is TC substance abuse treatment or the supportive residential setting. Typically, TC aftercare outcomes for prison TC graduates are compared to aftercare-as-usual, which can range across a wide variety of interventions. Few if any comparison groups have included a residential setting that emphasizes socialization and abstinence from drugs and alcohol - a hallmark of TC aftercare settings. This study proposes to compare the relative effectiveness of TC aftercare to an aftercare alternative that provides a supportive living environment without the professional treatment of TC aftercare. Oxford Houses (OH) provide, like TCs, a residential post-release setting that emphasizes socialization and abstinence from drugs and alcohol, but they do not include the formal therapeutic change interventions common to TCs, nor do they include any on-site access to drug abuse or health care professionals. Such a comparison will possibly clarify the value added of TC aftercare intervention processes not present in OHs.

The aims of this project are important from a public health perspective as there may be treatment matching, case management, and financing factors that could be manipulated to enhance the cost-effectiveness of community-based substance abuse treatment for offenders leaving prison. It is possible that both TC and OH aftercare modalities increase abstinence social support, self-efficacy, and employment, which mediate reductions in drug use, reincarceration, and health problems, but overall benefits are likely to be greater for TCs because they employ professional services and empirically based behavioral strategies. However, OHs might have advantages compared to more traditional post-incarceration modalities (e.g., low costs). Bringing scientific methods to the examination of TCs and the OH community-based recovery models for addiction might help to identify the "active ingredients" of these recovery settings. The proposed study will utilize ex-offenders randomly assigned to either TCs, OHs, or usual care post-release settings, and examine program effects (i.e., substance use, criminal and health outcomes), and economic factors associated with these models. A research finding from a study that contrasts these different approaches has the potential to influence practice and inform policy.

Several theoretically based hypotheses include:

TCs and OHs in comparison to usual aftercare will have less substance use, less criminal recidivism, and better health outcomes. TCs are expected to have better outcomes than OHs on these measures, due to the professionally structured and inpatient nature of TC.

Factors related to the programs (i.e., abstinence social support, self-efficacy, employment) will mediate the differential outcomes. For example, due to the inpatient nature of TCs and the requirement for employment to remain in OH, OH residents are expected to have more employment and earnings during the first year. However, these differences are expected to converge at 18 and 24 months. Usual aftercare should reflect the lowest employment and earning relative to TC and OH for all time periods.

The long term post release outcomes will be moderated by gender, ethnicity, substance abuse (i.e., severity and typology), and in-prison treatment (i.e., in prison TC fidelity, days in prison TC).

Although outcomes overall are expected to be best for TC, followed by OH and usual aftercare, we expect the cost-benefit ratios to be most favorable for OH, followed by TC, with the lowest cost benefit ratio for usual aftercare.

ELIGIBILITY:
Inclusion Criteria:

* have completed substance abuse treatment program, or attended 12-step program
* willing to live in a democratic residential setting, and pay rent
* Released from a prison or jail in the last 6 months

Exclusion Criteria:

* current substance addict/abuser
* have previously lived in an Oxford House
* not planning to go back to their own home or home of a relative following treatment
* sex offender, fire setter

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2007-10; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Substance Use | 2 years from baseline

SECONDARY OUTCOMES:
Criminal Recidivism | 2 years from baseline
Health Status | 2 years from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Leonard A Jason, Ph.D., Principal Investigator — DePaul University; Dave Mueller, Ph.D., Study Director — DePaul University
Locations (1):
- DePaul University, Chicago, Illinois, United States